CLINICAL TRIAL: NCT02065635
Title: Investigation of Changes in the Levels of Exhaled NO and Eosinophil Blood Count in Patients Undergoing Thyroidectomy by Two Different Methods of General Anesthesia Maintenance
Brief Title: Effect of Type of General Anesthesia Maintenance on Exhaled Nitric Oxide and Eosinophil Blood Count
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Associate Professor in Anesthesiology, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: NO-Artemis
Record Dates: First submitted 2014-02-15; First posted 2014-02-19 (Estimated); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Anesthesia; Exhaled Nitric Oxide; Eosinophil Blood Count
MeSH Terms: interventions — Maintenance; Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- maintenance with sevoflurane (Experimental): in patients allocated to the sevoflurane group, general anesthesia will be maintained with sevoflurane
  Interventions: Procedure: maintenance with sevoflurane
- maintenance with propofol (Active Comparator): in patients allocated to the propofol group, general anesthesia will be maintained with propofol
  Interventions: Procedure: maintenance with propofol

INTERVENTIONS:
Procedure: maintenance with sevoflurane — in patients allocated to the sevoflurane group, general anesthesia will be maintained with sevoflurane
  Arms: maintenance with sevoflurane
Procedure: maintenance with propofol — in patients allocated to the propofol group, general anesthesia will be maintained with propofol
  Arms: maintenance with propofol

SUMMARY:
* Nitric oxide (NO) is a free radical in gas state which plays an important role in a variety of processes relevant to respiratory physiology. It represents a means of detecting airway hyperresponsiveness and appears to have a strong correlation with the eosinophilic infiltration of the airway. Patients who suffered bronchospasm or laryngospasm intraoperatively or postoperatively showed higher levels of exhaled NO.
* Propofol modifies NO production by stimulating the constitutive synthesis of NO and by inhibiting the inducible production of NO. It seems to exert protective effects on acute lung injury (ALI) in experimental models and it can possibly reduce exhaled NO. There is also evidence that some intravenous anesthetic agents can influence chemotaxis of eosinophils in vitro.
* Variation of exhaled NO and eosinophils in surgical patients undergoing anesthesia has not been studied before. Therefore, the aim of this study will be to investigate the differential impact of maintenance of general anesthesia with propofol versus maintenance with sevoflurane on exhaled NO and eosinophil blood count.

DETAILED DESCRIPTION:
* Nitric oxide (NO) is a free radical in gas state which plays an important role in a variety of processes relevant to respiratory physiology. NO is produced by several cellular types (epithelial, endothelial, neuronic, inflammatory cells) (Gaston B, et al, 1994), it represents a means of detecting airway hyperresponsiveness and appears to have a strong correlation with the eosinophilic infiltration of the airway (Warke TJ, et al, 2002). Patients who suffered bronchospasm or laryngospasm intraoperatively or postoperatively showed higher levels of exhaled NO (Saraiva-Romanholo BM, et al, 2009).
* Propofol modifies NO production by stimulating the constitutive synthesis of NO and by inhibiting the inducible production of NO (González-Correa JA, et al, 2008). It seems to exert protective effects on acute lung injury in experimental models (Chu CH, et al, 2007; Chen HJ, et al, 2008) and possibly reduces exhaled NO (Fijałkowska A, et al, 2012). There is also evidence that some intravenous anesthetic agents can influence chemotaxis of eosinophils in vitro (Krumholz W, et al, 1999)
* Variation of exhaled NO and eosinophils in surgical patients undergoing anesthesia has not been studied before. Therefore, the aim of this study will be to investigate the differential impact of maintenance of general anesthesia with propofol versus maintenance with sevoflurane on exhaled NO and eosinophil blood count.
* Patients with ASA score I-III who undergo thyroidectomy under general anaesthesia will participate in this study. Thyroidectomy has been chosen for the following reasons: a) there will be consistency in both the surgeon and the type of surgery and as a result manipulations and surgical stress will be similar for all patients and b) abdominal walls are not manipulated at all during thyroidectomy and therefore postoperative measurement of exhaled NO will be easier and painless for patients.
* Patients will be randomized to one of two groups: one group with general anesthesia maintenance based on an intravenous agent (propofol) and a second group with general anesthesia maintenance based on an inhalational agent (sevoflurane).
* When patients arrive in the operating room, standard monitoring will be applied and exhaled NO will be measured immediately before induction with the NObreath® device ( Antus B, et al, 2010, Pisi R, et al, 2010) and a blood sample will be taken for eosinophil count measurement.
* During the patients' stay in the PACU and when Aldrete score is ≥8, exhaled NO will be measured again and a second blood sample will be taken. Exhaled NO will be measured again 24 hours postoperatively.
* The clinical implications of this study lie in the fact that it may provide further information on the effects of anesthetics (intravenous and inhalational) on the physiology and pathophysiology of the respiratory system. In addition, new evidence may come to light about the relationship between intravenous and inhalational agents and NO production.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, American Society of Anesthesiologists (ASA) distribution I-III, scheduled for thyroidectomy

Exclusion Criteria:

* patients with history of airway hyperreactivity (asthma, bronchitis)
* patients with history of allergy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-05; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
change of exhaled nitric oxide from preoperative status to immediate postoperative status | preoperatively, immediately postoperatively

SECONDARY OUTCOMES:
change of exhaled nitric oxide from preoperative status to 24 hours postoperatively | preoperatively, 24 hours postoperatively
change of eosinophil blood count from preoperative status to immediate postoperative status | preoperatively, immediately postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, PhD, DEAA, Principal Investigator — Aretaieion University Hospital; Artemis Vekrakou, MD, Principal Investigator — Aretaieion University Hospital; Eriphylli Argyra, PhD, Study Chair — Aretaieion University Hospital
Locations (1):
- Aretaieion University Hospital, Athens, Greece

REFERENCES:
- [Background] Gaston B, Drazen JM, Loscalzo J, Stamler JS. The biology of nitrogen oxides in the airways. Am J Respir Crit Care Med. 1994 Feb;149(2 Pt 1):538-51. doi: 10.1164/ajrccm.149.2.7508323.
- [Background] Warke TJ, Fitch PS, Brown V, Taylor R, Lyons JD, Ennis M, Shields MD. Exhaled nitric oxide correlates with airway eosinophils in childhood asthma. Thorax. 2002 May;57(5):383-7. doi: 10.1136/thorax.57.5.383. PMID 11978911
- [Background] Saraiva-Romanholo BM, Machado FS, Almeida FM, Nunes Mdo P, Martins MA, Vieira JE. Non-asthmatic patients show increased exhaled nitric oxide concentrations. Clinics (Sao Paulo). 2009;64(1):5-10. doi: 10.1590/s1807-59322009000100002. PMID 19142544
- [Background] Gonzalez-Correa JA, Cruz-Andreotti E, Arrebola MM, Lopez-Villodres JA, Jodar M, De La Cruz JP. Effects of propofol on the leukocyte nitric oxide pathway: in vitro and ex vivo studies in surgical patients. Naunyn Schmiedebergs Arch Pharmacol. 2008 Jan;376(5):331-9. doi: 10.1007/s00210-007-0220-4. Epub 2007 Dec 7. PMID 18064439
- [Background] Chu CH, David Liu D, Hsu YH, Lee KC, Chen HI. Propofol exerts protective effects on the acute lung injury induced by endotoxin in rats. Pulm Pharmacol Ther. 2007;20(5):503-12. doi: 10.1016/j.pupt.2006.03.006. Epub 2006 Apr 21. PMID 16713316
- [Background] Chen HI, Hsieh NK, Kao SJ, Su CF. Protective effects of propofol on acute lung injury induced by oleic acid in conscious rats. Crit Care Med. 2008 Apr;36(4):1214-21. doi: 10.1097/CCM.0b013e31816a0607. PMID 18379248
- [Background] Krumholz W, Abdulle O, Knecht J, Hempelmann G. Effects of i.v. anaesthetic agents on the chemotaxis of eosinophils in vitro. Br J Anaesth. 1999 Aug;83(2):333-5. doi: 10.1093/bja/83.2.333. PMID 10618953
- [Background] Antus B, Horvath I, Barta I. Assessment of exhaled nitric oxide by a new hand-held device. Respir Med. 2010 Sep;104(9):1377-80. doi: 10.1016/j.rmed.2010.06.005. Epub 2010 Jul 2. PMID 20594818
- [Background] Pisi R, Aiello M, Tzani P, Marangio E, Olivieri D, Chetta A. Measurement of fractional exhaled nitric oxide by a new portable device: comparison with the standard technique. J Asthma. 2010 Sep;47(7):805-9. doi: 10.3109/02770903.2010.485667. PMID 20670207
- See also: video about the use of NOBreath device — http://www.youtube.com/watch?v=ibHmStcBCtQ&feature=youtu.be
- See also: information about NOBreath device — http://www.bedfont.com/nobreath